CLINICAL TRIAL: NCT01895582
Title: Mycobacterium Tuberculosis Infection Diagnosis in Patients Above 75 Years Old/ Performance of Interferon Gamma Releasing Assays (IGRA)
Brief Title: Performance of IGRAs for TB Infection Diagnosis in Elderly
Acronym: IGRage
Status: Terminated | Type: Observational
Why Stopped: lack of recruitment of participants
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P110131; 2012-A00326-37 (Other: ANSM)
Record Dates: First submitted 2013-06-27; First posted 2013-07-10 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Ageing; Tuberculosis
Keywords: Ageing; Tuberculosis; Interferon gamma releasing tests
MeSH Terms: conditions — Tuberculosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Active TB-infected patients: TB-infected patients with bacteriological and histological evidences
  Interventions: Other: Blood samples
- Non active TB-infected patients (already met TB): some of elders have already met M tuberculosis before active antibiotherapy exists
  Interventions: Other: Blood samples
- Non active TB-infected patients (other diagnosis): same symptoms than two others groups but an other diagnosis
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — 4 blood tubes of lithium heparinate (5ml) 3 blood tubes of QTF-G-IT (1ml)
  1 blood dry tube (5ml)

SUMMARY:
Background: Diagnosis and screening for latent tuberculosis in old patients is of special interest in regards of the morbidity-mortality of this disease in that context.

TB-infection diagnosis based on immunological memory detection can be impaired with age. New blood tests (QFTB-G and T-SPOT.TB) specific for MTB infection have not been evaluated in those old patients.The primary endpoint of this study is the evaluation of the IGRAS for active TB diagnosis in patients above 75 years old.

DETAILED DESCRIPTION:
In vitro Interferon Gamma releasing Assay (IGRA) are recommended for LTBI screening as or instead of TST, but there accuracy in those old patients are not known: as immune responses are impaired in elderly and some of them have already met M tuberculosis before active antibiotherapy exists.The aim of this study is to evaluate characteristics of the two commercials tests IGRA T-spot-TB® and Quantiferon-TB-gold- in tube® and TST in old patients with or without active Tuberculosis.

Principal outcome:

- 3 tests performance for active TB diagnosis in patients older than 75 years-old

Secondary outcomes :

* concordance between IGRAs.
* non-concordant results analysis
* concordance of IGRAs results with time of TB-infection
* biobank

Methodology :Diagnostic test performance study

ELIGIBILITY:
Inclusion Criteria:

* Age > 75 years
* Consent signed
* hospitalized patient with start treatment of Tuberculosis disease
* French social right

Exclusion Criteria:

* Tuberculosis disease treatment since 7 days
* No 3 months follow-up possible
* Immunosuppression

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with suspected tuberculosis disease
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2013-07-17 (Actual); Primary Completion 2019-03-17 (Actual); Study Completion 2019-03-17 (Actual)

PRIMARY OUTCOMES:
Number of positive, indeterminate, negative tests in each group | month27

SECONDARY OUTCOMES:
Test results in clinical LTBI patients | month 27
Correlation with TB-infection date | month 27
  Test results (positive/negative) according to LTBI date
Blood samples collection in order to test new hypothesis in patients with non-concordant results | month 27
Performance comparison between tests (T-SPOT.TB®, Quantiferon-Gold-IT®) | month 27

CONTACTS AND LOCATIONS:
Overall Officials: Guislaine CARCELAIN, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Service de médecine interne, Bondy
  - Servive de Médecine Interne (Pr S. Herson), Paris
  - Service de Médecine Interne, Diabete et Maladies Métaboliques, Strasbourg